CLINICAL TRIAL: NCT06556940
Title: A Clinical Trial to Assess the Intraluminal Pharmacokinetics of LMN-401 in Individuals With Ileostomies
Brief Title: G.I. Pharmacokinetics of LMN-401 in Individuals With Ileostomies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lumen Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TD01
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Travelers Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Fast dissolving, uncoated LMN-401 tablets.
  Interventions: Biological: LMN-401
- Group 2 (Experimental): Slow dissolving, uncoated LMN-401 tablets.
  Interventions: Biological: LMN-401
- Group 3 (Experimental): Fast dissolving, enterically coated LMN-401 tablets.
  Interventions: Biological: LMN-401
- Group 4 (Experimental): Slow dissolving, enterically coated LMN-401 tablets.
  Interventions: Biological: LMN-401

INTERVENTIONS:
Biological: LMN-401 — Orally delivered tablets and capsules

SUMMARY:
The goal of this interventional study is to learn about the intraluminal pharmacokinetics (PK) of the investigational drug LMN-401 in adult healthy volunteers with ileostomies. LMN-401 is being developed as a potential new treatment for Traveler's Diarrhea. The study will also learn about the safety of the investigational drug LMN-401.

The main questions it aims to answer are:

* What is the timing and amount of components of investigational drug LMN-401 detected in the collected ileostomy material?
* Is LMN-401 safe and well tolerated in healthy volunteers taking the investigational drug?

Researchers will compare the timing and amount of investigational drug components detected in the ileostomy material in volunteers taking the investigational drug LMN-401 formulated into tablets with different properties. The impact of the study participant's fed or fasted state on the timing and amount of drug components detected in the ileostomy material will also be evaluated.

Each study participant will come into the research clinic for four study visits. Study participants will receive the investigational product formulated into tablets with different properties. Ileostomy material will be collected at baseline (pre-dose) and every two hours after investigational product dose administration for 10 hours.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 years and above
* Medically stable
* Mature and stable ileostomy (no revisions in past 6 months)
* Willing and able to participate in all study visits
* Willing and able to provide informed consent

Exclusion Criteria:

* Unable or unwilling to provide adequate informed consent
* Gastroparesis
* Using or planning to use anti-diarrheal medication
* Using or planning to use opioids
* Clinically significant disease
* Women who are pregnant, intending to become pregnant, or breastfeeding
* Non-English speakers

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-10-02 (Estimated); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Quantification of LMN-401 components in ileostomy material over time. | Ten hours post administration of study drug
  Measurement of individual VHH levels in ileostomy material over time after oral administration of LMN-401

CONTACTS AND LOCATIONS:
Locations (1):
- Coastal Digestive Health Research Institute Pty Ltd, Maroochydore, Australia